CLINICAL TRIAL: NCT03736577
Title: Psychotropic Drug Use in the Elderly Living in Nursing Homes - Associations With Clinical Symptoms and the Influence of a Structured Drug Review
Brief Title: Psychotropic Drug Use in the Elderly Living in Nursing Homes and the Influence of a Structured Drug Review
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Sykehuset Innlandet HF (Other); The Dam Foundation (Other); Norwegian Health Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Drug_review_nursing_homes
Record Dates: First submitted 2018-11-06; First posted 2018-11-09 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2020-09

CONDITIONS: Cognitive Symptom; Depression; Anxiety; Neuropsychiatric Syndrome; Quality of Life; Activity of Daily Living; Physical Health; Drug Use
MeSH Terms: conditions — Neurobehavioral Manifestations; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Two-armed cluster randomized trial. As the intervention is to introduce a new way to do drug chart reviews, to prevent contamination bias within the nursing home the whole nursing home will have to be treated as a cluster. The recruited nursing homes will be randomized by a statistician to either intervention or control. Before randomization, both physicians working in the recruited facilities and selected personnel, i.e. specialized nurses, will attend a three hours lecture on dementia, depression and anxiety and psychosis on the elderly.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NorGeP-NH (Experimental): Initially, a three hours lecture on dementia, depression, anxiety and psychosis on the elderly will be held. Both physicians working in the facilities and selected personnel, i.e. specialized nurses, will attend.
  Intervention: Drug reviews with NorGeP-NH Physicians in the intervention group will attend a 1-2 hours lecture about psychopharmacology and drug review. They will learn how to do drug reviews with the Norwegian general practice criteria - Nursing homes (NorGeP-NH) and they will do a structured drug review on the participants' drug charts.
  Interventions: Other: Drug reviews with NorGeP-NH
- Control nursing home (No Intervention): Initially, a three hours lecture on dementia, depression, anxiety and psychosis on the elderly will be held. Both physicians working in the facilities and selected personnel, i.e. specialized nurses, will attend. Physicians will not attend any lecture about drug reviews and they will keep treating participants "as usual".

INTERVENTIONS:
Other: Drug reviews with NorGeP-NH — Physicians in the intervention group will attend a 1-2 hours lecture about psychopharmacology and drug review. They will learn how to do drug reviews with the Norwegian general practice criteria - Nursing homes (NorGeP-NH). The nursing home physicians will do the drug review on the participants' drug charts
  Arms: NorGeP-NH

SUMMARY:
The overall aim of this study is to explore if a structured drug review will change clinical symptoms and the psychotropic drugs prescription rate in the elderly living in nursing homes (participants of the study). The study will examine how training of nursing home physicians on reviewing prescription lists using the Norwegian general practice criteria - Nursing homes (NorGeP-NH) will influence the participants' clinical symptoms such as cognition, depression, anxiety and their quality of life. Secondary, we will analyse how a structured drug review will influence further psychotropic drug prescribing rates in nursing homes.

The hypothesis for this study are:

1. Training of nursing home physicians on doing a systematic drug review will decrease the participants' clinical symptoms and improve their Quality of Life.
2. A systematic drug review will decrease the psychotropic drug prescription rates compared to before the drug review.

DETAILED DESCRIPTION:
Norwegian national guidelines recommend a very cautious use of psychotropic drugs in the elderly, especially for treating dementia-related symptoms. These drugs should be used at a very low dosage and for as short a time as possible. Despite these strict guidelines, patients with and without dementia living in nursing homes still receive a high amount of psychotropic drugs. Thus, there should be a higher focus on lowering the use of psychotropic medications in nursing homes. A reduction of prescription of potential harmful and inappropriate drugs for the elderly may improve the clinical symptoms of the patients, reduce the interaction between drugs and the side-effects, and thereby improving the quality of life of the patients.

In 2018 the Norwegian Institute of Public Health updated a report about the general health in the Norwegian elderly population. This report shows that prescription rates for the majority of drugs in the population above 65 years of age have increased in the past 11 years. Unfortunately, Norway does not have a prescription registry for patients living in nursing homes and according to the same report the drug use and the increase of prescription rates in nursing homes is underestimated. During the last years Norwegian authorities, media and user organizations have shown a particular interest in this subject, showing how clinical practice still differs from national and international guidelines, and focusing on the severity of polypharmacy in the elderly living in institutions, particularly concerning patients with dementia receiving psychotropic drugs.

As a result of missing data concerning the real use and increase of drug prescriptions in nursing homes, our study will keep exploring the psychotropic drug use in the elderly population living in Norwegian nursing homes, and it will increase the knowledge about risk factors associated to higher prescription rates. The effect of structured reviews with NorGeP is understudied, and the proposed randomized controlled trial could therefore add valuable knowledge to the field, by exploring how specific training for health personnel working in nursing homes will affect drug prescription in the future.

ELIGIBILITY:
Inclusion Criteria:

* The participant is living in a participating nursing home
* Expected stay for more than 12 weeks

Exclusion Criteria:

* Severe somatic or psychiatric disease where the participant is too debilitated or not able to cooperate, or where the examination or assessment would cause a too big psychological and physical burden (i.e. severe psychotic state)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life: QUALID | 12 weeks
  Quality of Life in Late-Stage Dementia (QUALID) - Reporting the QoL of the patients on a scale from 11-55 where lower score indicates better QoL

SECONDARY OUTCOMES:
Number of drugs prescribed | 8 weeks
  Registration with Anatomical Therapeutic Chemical (ATC) code and daily dosage
Number of drugs prescribed | 12 weeks
  Registration with ATC code and daily dosage
Depression | 8 weeks
  Cornell Scale for depression in dementia (CDSS). Score range 0-38. A score totaling six (6) or less indicates no depression. A score totaling between seven (7) and eleven (11) indicates possible depression. A score totaling twelve (12) or more indicates major depression.
Depression | 12 weeks
  Cornell Scale for depression in dementia (CDSS). Score range 0-38. A score totaling six (6) or less indicates no depression. A score totaling between seven (7) and eleven (11) indicates possible depression. A score totaling twelve (12) or more indicates major depression.
Depression | 8 weeks
  Montgomery and Åsberg Depression Rating Scale (MADRS). Score range 0-60. A score totaling six (6) or less indicate no depression. A score totaling between seven (7) and nineteen (19) indicates mild depression. A score totaling between twenty (20) and thirty-four (34) indicates moderate depression. A score totaling thirty-five (35) or more indicates severe depression.
Depression | 12 weeks
  Montgomery and Åsberg Depression Rating Scale (MADRS). Score range 0-60. A score totaling six (6) or less indicate no depression. A score totaling between seven (7) and nineteen (19) indicates mild depression. A score totaling between twenty (20) and thirty-four (34) indicates moderate depression. A score totaling thirty-five (35) or more indicates severe depression.
Neuropsychiatric symptoms - agitation | 8 weeks
  Neuropsychiatric Inventory - agitation subsyndrome. Instrument used to evaluate the presence and severity of neuropsychiatric symptoms
Neuropsychiatric symptoms - agitation | 12 weeks
  Neuropsychiatric Inventory - agitation subsyndrome. Instrument used to evaluate the presence and severity of neuropsychiatric symptoms
Neuropsychiatric symptoms - affective symptoms | 8 weeks
  Neuropsychiatric Inventory - affective subsyndrome. Instrument used to evaluate the presence and severity of neuropsychiatric symptoms
Neuropsychiatric symptoms - affective symptoms | 12 weeks
  Neuropsychiatric Inventory - affective subsyndrome. Instrument used to evaluate the presence and severity of neuropsychiatric symptoms
Cognition | 8 weeks
  Montreal Cognitive Assessment. Score range 0-30. A score totaling twenty-six (26) or more indicates no cognitive impairment. A score totaling twenty-five (25) or less indicates cognitive impairment.
Cognition | 12 weeks
  Montreal Cognitive Assessment. Score range 0-30. A score totaling twenty-six (26) or more indicates no cognitive impairment. A score totaling twenty-five (25) or less indicates cognitive impairment.
Cognition | 8 weeks
  Clinical Dementia Rating Scale. The total score is calculated through a particular scoring algorithm. The final score can result in the following values: 0 = normal; 0,5 = very mild dementia; 1 = mild dementia; 2 = moderate dementia; 3 = severe dementia
Cognition | 12 weeks
  Clinical Dementia Rating Scale. The total score is calculated through a particular scoring algorithm. The final score can result in the following values: 0 = normal; 0,5 = very mild dementia; 1 = mild dementia; 2 = moderate dementia; 3 = severe dementia
Anxiety | 8 weeks
  Geriatric Anxiety Inventory - a 20-items instrument to evaluate the severity of anxiety. Score range 0 - 20. A higher score indicates a higher severity of anxiety.
Anxiety | 12 weeks
  Geriatric Anxiety Inventory - a 20-items instrument to evaluate the severity of anxiety. Score range 0 - 20. A higher score indicates a higher severity of anxiety.
Activity of daily living | 8 weeks
  Physical Self-Maintenance Scale. A 6-items instrument to describe a person's highest level of functioning. Each item can be scored from 1 to 5. A lower score indicates better functioning.
Activity of daily living | 12 weeks
  Physical Self-Maintenance Scale. A 6-items instrument to describe a person's highest level of functioning. Each item can be scored from 1 to 5. A lower score indicates better functioning.
Physical health | Participants will be assessed at baseline, after 8 weeks and 12 weeks
  General Medical Health Rating
Physical health | Participants will be assessed at baseline, after 8 weeks and 12 weeks
  Charlson Comorbidity Index
Physical health | Participants will be assessed at baseline, after 8 weeks and 12 weeks
  The timed "up and go" test

CONTACTS AND LOCATIONS:
Overall Officials: Sverre Bergh, MD, PhD, Principal Investigator — Innlandet Hospital Trust, Postboks 104, 2381 Brumunddal, Norway
Locations (1):
- Østfold Hospital Trust - Dept. of mental health, Grålum, Norway

IPD SHARING:
Plan to Share IPD: Yes
Upon request, and after approval by the Regional committee for medical and health research ethics, IPD that underlie results in a publication might be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Starting 6 months after results publication.
Access Criteria: Because of the sensitive nature of the data, any access request will have to be submitted to the Central Contact Person and / or Central Contact Backup. After a preliminary review, the request will be forwarded to Regional committee for medical and health research ethics for approval.

REFERENCES:
- [Background] Nyborg G, Straand J, Klovning A, Brekke M. The Norwegian General Practice--Nursing Home criteria (NORGEP-NH) for potentially inappropriate medication use: A web-based Delphi study. Scand J Prim Health Care. 2015 Jun;33(2):134-41. doi: 10.3109/02813432.2015.1041833. Epub 2015 Jun 23. PMID 26100966
- [Background] Nyborg G, Brekke M, Straand J, Gjelstad S, Romoren M. Potentially inappropriate medication use in nursing homes: an observational study using the NORGEP-NH criteria. BMC Geriatr. 2017 Sep 19;17(1):220. doi: 10.1186/s12877-017-0608-z. PMID 28927372
- See also: Report from the Norwegian Institute of Public Health — https://www.fhi.no/nettpub/hin/grupper/eldre/
- See also: Norwegian national guidelines on dementia — https://helsedirektoratet.no/retningslinjer/nasjonal-faglig-retningslinje-om-demens